CLINICAL TRIAL: NCT02646891
Title: Phase I/II Double-blind, Randomized, Placebo-controlled, Descending Age, Dose-escalation Study of the Safety, and Immunogenicity of the Trivalent P2-VP8 Subunit Rotavirus Vaccine in Healthy South African Adults, Toddlers and Infants
Brief Title: Safety and Immunogenicity Study of Trivalent P2-VP8 Subunit Rotavirus Vaccine in Adults, Toddlers and Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-041
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: Rotavirus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Adults: Placebo (Placebo Comparator): Adults received three intramuscular injections of placebo four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Placebo
- Adults: 30 µg P2-VP8 (Experimental): Adults received three intramuscular injections of 30 µg trivalent P2-VP8 subunit rotavirus vaccine four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine
- Adults: 90 µg P2-VP8 (Experimental): Adults received three intramuscular injections of 90 µg trivalent P2-VP8 subunit rotavirus vaccine four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine
- Toddlers: Placebo (Placebo Comparator): Toddlers received one intramuscular injection of placebo on Day 0.
  Interventions: Biological: Placebo
- Toddlers: 30 µg P2-VP8 (Experimental): Toddlers received one intramuscular injection of 30 µg trivalent P2-VP8 subunit rotavirus vaccine on Day 0.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine
- Toddlers: 90 µg P2-VP8 (Experimental): Toddlers received one intramuscular injection of 90 µg trivalent P2-VP8 subunit rotavirus vaccine on Day 0.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine
- Infants: Placebo (Placebo Comparator): Infants received three intramuscular injections of placebo four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Placebo
- Infants: 15 µg P2-VP8 (Experimental): Infants received three intramuscular injections of 15 µg trivalent P2-VP8 subunit rotavirus vaccine four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine
- Infants: 30 µg P2-VP8 (Experimental): Infants received three intramuscular injections of 30 µg trivalent P2-VP8 subunit rotavirus vaccine four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine
- Infants: 90 µg P2-VP8 (Experimental): Infants received three intramuscular injections of 90 µg trivalent P2-VP8 subunit rotavirus vaccine four weeks apart on Days 0, 28, and 56.
  Interventions: Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine

INTERVENTIONS:
Biological: Trivalent P2-VP8 Subunit Rotavirus Vaccine — Manufactured and supplied by the Walter Reed Army Institute of Research (WRAIR) Pilot Bioproduction Facility (BPF). The trivalent P2-VP8 vaccine was formulated as a sterile suspension containing a total of 360 µg of protein (120 µg of each P type) per mL adsorbed to aluminum hydroxide (1.125 mg of aluminum per mL in a phosphate buffer, pH 7).
  Arms: Adults: 30 µg P2-VP8; Adults: 90 µg P2-VP8; Infants: 15 µg P2-VP8; Infants: 30 µg P2-VP8; Infants: 90 µg P2-VP8; Toddlers: 30 µg P2-VP8; Toddlers: 90 µg P2-VP8
Biological: Placebo — Sodium Chloride 0.9%, USP for Injection
  Arms: Adults: Placebo; Infants: Placebo; Toddlers: Placebo

SUMMARY:
This is is a study of a parenteral trivalent rotavirus vaccine (P2-VP8 subunit rotavirus vaccine). The study examined the safety and immunogenicity of three dose levels of this vaccine in healthy South African adults, toddlers and infants. Progression from one dose level to another and to the next age group population was based on the assessment of safety information from the lowest dose and older age group.

The primary safety hypothesis is that the P2-VP8 subunit rotavirus vaccine is safe and well-tolerated. The primary immunogenicity hypothesis is that the trivalent P2-VP8 subunit rotavirus vaccine is immunogenic in infant participants and will induce an immune response to at least 2 of the 3 strains in 60% or more of participants in at least one of the study groups.

DETAILED DESCRIPTION:
The P2-VP8 vaccine tested in this study was developed by Dr. Taka Hoshino at National Institute of Allergy and Infectious Diseases (NIAID). The monovalent (P[8]) vaccine previously tested consisted of bacteria-expressed VP8 subunit from the Wa strain of human rotaviruses (G1[P8]). A deoxyribonucleic acid (DNA) segment encoding the sequence of P2 epitope from tetanus toxin was fused to the VP8 sequence, resulting in this chimeric protein vaccine (P2-VP8). Dr. Hoshino's laboratory demonstrated in preclinical testing that the immunogenicity of these VP8 proteins could be significantly enhanced when fused with the P2 epitope of tetanus toxin, which exerts a strong T cell helper function. Further, immunization of neonatal piglets with a P2-VP8-P[8] chimeric protein conferred significant protection against experimental rotavirus gastroenteritis. Based on results of the initial first-in-human testing of the monovalent (P[8]) vaccine, a trivalent vaccine that includes antigens from P[4], P[6] and P[8] strains (DS-1, 1076 and Wa, respectively) has been developed to broaden responses for these 3 P-types, which together are responsible for the vast majority of global disease burden. The trivalent vaccine was assessed in this study.

The first clinical testing of the monovalent (P[8]) P2-VP8 subunit rotavirus vaccine was performed in 18-45 year old adults in North America. Overall, the vaccine was well-tolerated at all three dose levels, was associated with only mild transient local reactogenicity, and no safety concerns were identified. Almost all vaccine recipients demonstrated greater than 4-fold rise in IgG and IgA response to P2-VP8 antigen by enzyme-linked immunosorbent assay (ELISA) after three vaccinations: only one vaccine recipient did not demonstrate an immunoglobulin G (IgG) response (in the 30 µg group) and all vaccine recipients demonstrated immunoglobulin A (IgA) responses. Neutralizing antibody responses were also encouraging, with clear increases in geometric mean titers (GMTs) for all three dose levels at one month post-third study injection (Day 84) compared to pre-vaccination levels. Neutralizing antibody responses to heterologous rotavirus strains were most robust to P[8] strains, moderate to the P[4] strain and fairly limited to the P[6] strain.

Clinical testing of the monovalent (P[8]) P2-VP8 subunit rotavirus vaccine was initiated in South African toddlers and infants in 2014. The vaccine was generally well-tolerated at all three dose levels. In both toddlers and infants, when local reactogenicity was reported, it was transient, rarely greater than mild, and never severe. When present, systemic reactogenicity was also transient and generally mild, without discernable dose effect. In the dose-escalation phase of the testing in the infant cohorts, the study injections were paused temporarily due to findings of severe neutropenia on post-vaccination laboratory monitoring in three participants (two infants and one toddler) but were later resumed after the Safety Review Committee assessed that the data did not support relation to the study vaccine. The primary serology results in the infant cohorts were close to universal responses, with substantial increases in titer as demonstrated by mean-fold increase in GMT. In infants receiving the 30 µg dose, the GMT rose from a baseline value of 107 to a post-vaccination value of 9,583. Although not as dramatic as the IgG responses, there were good IgA responses to P2-VP8, with the seroresponse rate over 80% in infants receiving 30 µg of vaccine. The 60 µg dose did not appear to provide any better response than the 30 µg dose, although this study was not powered for that comparison.

In summary, the P2-VP8 monovalent vaccine was generally well-tolerated in healthy South African infants, and there was no evidence that the higher vaccine dose (60 µg) provided any benefit in serologic responses or impact on shedding of Rotarix compared to the lower dose (30 µg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (≥ 18 and ≤ 45 years), toddlers (≥ 2 and ≤ 3 years), and infants (≥ 6 and ≤ 8 weeks)
* Participants will remain in the area during the study
* Females of childbearing potential must not be pregnant or breastfeeding, and willing to use adequate method of contraception during the trial.

Exclusion Criteria:

* Presence of fever or other acute illness
* concurrent participation in another clinical trial
* Presence of malnutrition or other systemic disorder.
* Infants with history of premature birth (< 37 week gestational age)
* History of congenital abdominal disorders or surgery
* Suspected or known impairment of immune function
* Infants who have received rotavirus vaccine in the past
* Known sensitivity to any components of the vaccine
* History of anaphylactic reaction
* Major congenital or genetic defect
* Unwillingness to follow study schedule
* Receipt of immunoglobulin therapy or blood products in last 6 months
* History of chronic immunosuppressive medications (with the exception of inhaled or topical steroids)
* Any medical condition that, in the judgement of the investigator, would interfere with the protocol, or would interfere with participant's ability to adhere to the study protocol.
* Clinically significant screening laboratory value
* Human immunodeficiency virus (HIV) infection

Ages: 6 Weeks to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 618 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Groom, MBBCh, Study Chair — Chris Hani Baragwanath Hospital
Locations (3):
- South Africa (3):
  - Respiratory and Meningeal Pathogens Research Unit (RMPRU), Johannesburg, Gauteng
  - Shandukani Research Centre, Johannesburg
  - Family Clinical Research Unit (FAM-CRU) Stellenbosch Univ, Stellenbosch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groome MJ, Fairlie L, Morrison J, Fix A, Koen A, Masenya M, Jose L, Madhi SA, Page N, McNeal M, Dally L, Cho I, Power M, Flores J, Cryz S. Safety and immunogenicity of a parenteral trivalent P2-VP8 subunit rotavirus vaccine: a multisite, randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2020 Jul;20(7):851-863. doi: 10.1016/S1473-3099(20)30001-3. Epub 2020 Apr 3. PMID 32251641

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult: Placebo: Adult participants who received three intramuscular injections of placebo four weeks apart on days 0, 28, and 56. Approximately half of the participants were compared to the arm receiving the 30 µg dose of P2-VP8; once the safety of this dose was established, the other half were compared to the arm receiving 90 µg.
- Adult: P2-VP8 (30 µg): Adult participants who received three intramuscular injections of Trivalent P2-VP8 Subunit Rotavirus Vaccine (30 µg) four weeks apart on days 0, 28, and 56.
- Adult: P2-VP8 (90 µg): Adult participants who received three intramuscular injections of Trivalent P2-VP8 Subunit Rotavirus Vaccine (90 µg) four weeks apart on days 0, 28, and 56.
- Toddler: Placebo: Toddler participants who received one intramuscular injection of placebo on day 0. Approximately half of the participants were compared to the arm receiving the 30 µg dose of P2-VP8; once the safety of this dose was established, the other half were compared to the arm receiving 90 µg.
- Toddler: P2-VP8 (30 µg): Toddler participants who received one intramuscular injections of Trivalent P2-VP8 Subunit Rotavirus Vaccine (30 µg) on day 0.
- Toddler: P2-VP8 (90 µg): Toddler participants who received one intramuscular injection of Trivalent P2-VP8 Subunit Rotavirus Vaccine (90 µg) on day 0.
- Infant: Placebo: Infant participants who received three intramuscular injections of placebo four weeks apart on days 0, 28, and 56. Approximately one third of the participants were compared to the arm receiving the 15 µg dose of P2-VP8; once the safety of the 15 µg dose was established, one third of the participants were compared to the arm receiving 30 µg; and the last third were compared to the arm receiving 90 µg after the safety of the 30 µg dose was established.
- Infant: P2-VP8 (15 µg): Infant participants who received three intramuscular injections of Trivalent P2-VP8 Subunit Rotavirus Vaccine (15 µg) four weeks apart on days 0, 28, and 56.
- Infant: P2-VP8 (30 µg): Infant participants who received three intramuscular injections of Trivalent P2-VP8 Subunit Rotavirus Vaccine (30 µg) four weeks apart on days 0, 28, and 56.
- Infant: P2-VP8 (90 µg): Infant participants who received three intramuscular injections of Trivalent P2-VP8 Subunit Rotavirus Vaccine (90 µg) four weeks apart on days 0, 28, and 56.
Period: Overall Study
Arm/Group | Adult: Placebo | Adult: P2-VP8 (30 µg) | Adult: P2-VP8 (90 µg) | Toddler: Placebo | Toddler: P2-VP8 (30 µg) | Toddler: P2-VP8 (90 µg) | Infant: Placebo | Infant: P2-VP8 (15 µg) | Infant: P2-VP8 (30 µg) | Infant: P2-VP8 (90 µg)
Started | 6 | 12 | 12 | 6 | 12 | 12 | 139 | 140 | 140 | 139
Received at Least 1 Dose | 6 | 12 | 12 | 6 | 12 | 12 | 139 | 139 (One participant was randomized but determined to be ineligible pre-vaccination.) | 140 | 139
Completed | 4 | 11 | 11 | 6 | 12 | 12 | 130 | 127 | 130 | 134
Not Completed | 2 | 1 | 1 | 0 | 0 | 0 | 9 | 13 | 10 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 0 | 0 | 5 | 9 | 7 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8 | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8 | Total
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12 | 139 | 140 | 140 | 139 | 618
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (2.1) | 32.0 (4.8) | 26.0 (6.0) | 2.6 (0.1) | 2.6 (0.2) | 2.5 (0.2) | 0.13 (0.01) | 0.13 (0.01) | 0.13 (0.01) | 0.13 (0.01) | 16.3 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9 | 4 | 7 | 5 | 67 | 66 | 76 | 64 | 307
  Male | 3 | 6 | 3 | 2 | 5 | 7 | 72 | 74 | 64 | 75 | 311
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 6 | 12 | 12 | 6 | 12 | 12 | 137 | 138 | 138 | 136 | 609
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Colored | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 8
  Unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: centimeters] — Population: Height was not collected for one participant.
  centimeters
    number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12 | 138 | 140 | 140 | 139 | 617
    (all) | 167.0 (12.5) | 164.4 (10.6) | 160.6 (8.3) | 88.8 (6.8) | 86.4 (7.6) | 88.5 (4.3) | 55.4 (2.35) | 54.9 (2.48) | 55.1 (2.24) | 55.3 (1.98) | 62.0 (24.2)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Weight for one participant was missing.
  kilograms
    number analyzed (Participants) | 6 | 12 | 11 | 6 | 12 | 12 | 139 | 140 | 140 | 139 | 617
    (all) | 62.7 (8.1) | 68.7 (10.4) | 61.2 (10.2) | 13.8 (2.4) | 12.6 (1.5) | 13.5 (2.3) | 4.9 (0.59) | 4.8 (0.66) | 4.8 (0.54) | 4.9 (0.58) | 8.1 (13.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AE) Within 28 Days of Any Vaccination
Description: Any symptom starting after 7 days post any study injection was recorded as an adverse event. A serious adverse event (SAE) is any event that occurred from the first dose of study drug that resulted in any of the following outcomes:
  1. Death
  2. Life-threatening AE
  3. Inpatient hospitalization or prolongation of existing hospitalization
  4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  5. Congenital abnormality or birth defect
  6. Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant or require medical or surgical intervention to prevent one of the outcomes listed above.
  The severity of adverse events was graded from Mild (grade 1) to Life Threatening (grade 4).
  AEs related to study drug were those events for which there was a reasonable possibility that the study drug caused the event In the opinion of the site investigator.
Time Frame: Up to 28 days after any vaccination (up to Day 28 for toddlers and up to Day 84 for infants and adults)
Population: Safety population included all participants who were randomized and received at least one injection of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8 | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12 | 139 | 139 | 140 | 139
Participants
  Any serious adverse event | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 8 | 4 | 4
  Any AE | 2 | 8 | 9 | 3 | 8 | 6 | 119 | 118 | 122 | 124
  Any grade 2 or higher AE | 0 | 2 | 1 | 0 | 1 | 1 | 19 | 24 | 18 | 20
  Any AE related to study drug | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 3 | 2
  Any grade 2 or higher AE related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

2. Primary Outcome: Number of Participants With Local or Systemic Reactions Within 7 Day of Vaccination
Description: Reactogenicity data (solicited signs or symptoms) were assessed for 7 days after each injection. Participants and parents were instructed to assess and record daily local reactions (injection site pain/tenderness, redness, swelling, itching), as well as systemic signs and symptoms (fever, headache, vomiting, nausea, fatigue, chills and myalgia for adults; and fever, vomiting, decreased appetite, irritability, and decreased activity for toddlers and infants) in a participant memory aid. Reactions were graded on a scale from mild (Grade 1) to life-threatening (Grade 4).
  The overall number of participants who experienced any local or systemic reaction is reported. Grades are based on maximum severity per participant.
Time Frame: 7 days following each vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8 | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12 | 139 | 139 | 140 | 139
Participants
  Any local reaction | 1 | 7 | 9 | 2 | 6 | 2 | 93 | 102 | 109 | 108
  Local reaction: Grade 1 | 1 | 6 | 6 | 2 | 4 | 2 | 84 | 83 | 96 | 92
  Local reaction: Grade 2 | 0 | 1 | 3 | 0 | 2 | 0 | 9 | 19 | 13 | 16
  Local reaction: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Local reaction: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any systemic reaction | 5 | 6 | 9 | 4 | 5 | 2 | 116 | 114 | 113 | 115
  Systemic reaction: Grade 1 | 5 | 6 | 6 | 3 | 5 | 2 | 86 | 70 | 83 | 73
  Systemic reaction : Grade 2 | 0 | 0 | 3 | 1 | 0 | 0 | 30 | 39 | 28 | 40
  Systemic reaction: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2
  Systemic reaction: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Infants With Anti-P2-VP8 Immunoglobulin G (IgG) Seroresponse 4 Weeks After the Third Vaccination, by Vaccine Antigen
Description: Seroresponse was defined as a four-fold rise or greater in antibody titer between Baseline and 28 days after the third injection (Day 84). Measured by enzyme-linked immunosorbent assay (ELISA) and adjusted for decay in maternal IgG antibodies. The estimated maternal antibody half-life was derived from linear regression of Log2 transformed titers in placebo recipients from the combined infant cohorts.
Time Frame: Day 84
Population: Per-protocol population included all randomized participants who adhered to the protocol, completed all their scheduled visits and vaccinations up to the analysis time point and presented no major protocol violations (defined as a protocol violation that was considered to have an impact on the immunogenicity results of the study).
Measure: Count of Participants; unit: Participants
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 130 | 132 | 132 | 134
Participants
  P[4] | 16 | 131 | 130 | 134
  P[6] | 38 | 131 | 132 | 134
  P[8] | 13 | 131 | 130 | 134
  Any 2 antigens | 16 | 131 | 130 | 134
  All 3 antigens | 11 | 131 | 130 | 134

4. Primary Outcome: Number of Infants With Anti-P2-VP8 Immunoglobulin A (IgA) Seroresponse 4 Weeks After the Third Vaccination, by Vaccine Antigen
Description: Seroresponse was defined as a four-fold rise or greater in antibody titer between Baseline and 28 days after the final injection (Day 84). Measured by enzyme-linked immunosorbent assay (ELISA) to whole viral lysate.
Time Frame: Day 84
Population: Per-protocol population participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 130 | 131 | 132 | 134
Participants
  P[4]: number analyzed (Participants) | 130 | 130 | 132 | 134
  P[4] | 13 | 35 | 40 | 32
  P[6]: number analyzed (Participants) | 130 | 131 | 131 | 134
  P[6] | 13 | 37 | 44 | 34
  P[8]: number analyzed (Participants) | 130 | 129 | 130 | 131
  P[8] | 11 | 36 | 26 | 28
  Any 2 antigens: number analyzed (Participants) | 130 | 130 | 132 | 134
  Any 2 antigens | 11 | 34 | 35 | 29
  All 3 antigens: number analyzed (Participants) | 130 | 128 | 129 | 131
  All 3 antigens | 7 | 19 | 16 | 16

5. Primary Outcome: Number of Infants With Neutralizing Antibody Responses 4 Weeks After the Third Vaccination to Each Rotavirus Strain
Description: Neutralizing antibody response was defined as a ≥ 2.7-fold rise in antibody titer between Baseline and 28 days after the final injection (Day 84). Neutralizing antibodies to each of the three rotavirus strains from which the vaccine antigens were derived (Wa, DS-1, and 1076) were measured using a validated assay. For infants, antibody titer was adjusted for decay in maternal antibodies.
Time Frame: Day 84
Population: Per-protocol population participants with available data for each strain
Measure: Count of Participants; unit: Participants
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 130 | 132 | 132 | 134
Participants
  Rotavirus strain Wa | 26 | 96 | 107 | 105
  Rotavirus strain DS-1: number analyzed (Participants) | 130 | 131 | 132 | 134
  Rotavirus strain DS-1 | 26 | 100 | 105 | 108
  Rotavirus strain 1076 | 16 | 90 | 103 | 109
  Any 2 strains | 15 | 101 | 108 | 114
  All 3 strains: number analyzed (Participants) | 130 | 131 | 132 | 134
  All 3 strains | 10 | 65 | 81 | 83

6. Primary Outcome: Anti-P2-VP8 Immunoglobulin G (IgG) Geometric Mean Titers Among Infants, by Vaccine Antigen
Description: Measured by ELISA at Baseline, 28 days after the second injection (Day 56 pre-vaccination; secondary outcome) and 28 days after the third and final injection (Day 84; primary outcome).
Time Frame: Baseline and Days 56 (pre-vaccination) and 84
Population: Per-protocol population; participants with valid specimens at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Infants: Placebo; Infants: 15 µg P2-VP8: Infants received three intramuscular injections of 15 µg trivalent P2-VP8 subunit rotavirus vaccine four weeks apart on Days 0, 28, and 56.
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 135 | 137 | 132 | 137
titer
  P[4]: Baseline | 73 [57 to 94] | 80 [64 to 101] | 62 [48 to 79] | 76 [62 to 94]
  P[4]: Day 56: number analyzed (Participants) | 135 | 137 | 131 | 136
  P[4]: Day 56 | 30 [24 to 38] | 1456 [1244 to 1705] | 1849 [1581 to 2163] | 2424 [2099 to 2800]
  P[4]: Day 84: number analyzed (Participants) | 130 | 132 | 132 | 134
  P[4]: Day 84 | 28 [22 to 36] | 3888 [3313 to 4562] | 4205 [3692 to 4789] | 5244 [4729 to 5815]
  P[6]: Baseline | 67 [52 to 86] | 73 [58 to 92] | 63 [49 to 82] | 66 [52 to 83]
  P[6]: Day 56: number analyzed (Participants) | 135 | 137 | 131 | 136
  P[6]: Day 56 | 47 [38 to 58] | 5031 [4305 to 5880] | 5709 [4932 to 6609] | 7122 [6176 to 8213]
  P[6]: Day 84: number analyzed (Participants) | 130 | 132 | 132 | 134
  P[6]: Day 84 | 50 [39 to 64] | 14028 [11980 to 16426] | 14724 [13181 to 16447] | 17085 [15295 to 19085]
  P[8]: Baseline | 84 [66 to 109] | 86 [69 to 109] | 74 [59 to 94] | 81 [65 to 100]
  P[8]: Day 56: number analyzed (Participants) | 134 | 137 | 131 | 136
  P[8]: Day 56 | 35 [28 to 45] | 1897 [1616 to 2227] | 2323 [1985 to 2719] | 3050 [2621 to 3549]
  P[8]: Day 84: number analyzed (Participants) | 130 | 132 | 132 | 134
  P[8]: Day 84 | 30 [23 to 39] | 5365 [4454 to 6321] | 5792 [5086 to 6595] | 7088 [6314 to 7958]

7. Primary Outcome: Anti-P2-VP8 Immunoglobulin A (IgA) Geometric Mean Titers Among Infants, by Vaccine Antigen
Description: as for outcome 6
Time Frame: Baseline and Days 56 (pre-vaccination) and 84
Population: Per-protocol population; participants with valid specimens at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 135 | 137 | 132 | 137
titer
  P[4]: Baseline: number analyzed (Participants) | 135 | 136 | 132 | 137
  P[4]: Baseline | 5 [5 to 5] | 5 [5 to 6] | 5 [5 to 5] | 5 [5 to 5]
  P[4]: Day 56: number analyzed (Participants) | 134 | 136 | 131 | 136
  P[4]: Day 56 | 6 [5 to 7] | 9 [7 to 11] | 10 [8 to 12] | 9 [7 to 10]
  P[4]: Day 84: number analyzed (Participants) | 130 | 130 | 132 | 134
  P[4]: Day 84 | 7 [5 to 8] | 13 [10 to 17] | 12 [10 to 15] | 10 [9 to 12]
  P[6]: Baseline | 5 [4 to 5] | 5 [5 to 6] | 5 [4 to 5] | 5 [5 to 6]
  P[6]: Day 56: number analyzed (Participants) | 135 | 137 | 131 | 136
  P[6]: Day 56 | 6 [6 to 7] | 9 [7 to 10] | 10 [8 to 12] | 10 [8 to 12]
  P[6]: Day 84: number analyzed (Participants) | 130 | 131 | 131 | 134
  P[6]: Day 84 | 7 [6 to 8] | 12 [10 to 15] | 13 [10 to 15] | 12 [10 to 14]
  P[8]: Baseline: number analyzed (Participants) | 135 | 136 | 132 | 137
  P[8]: Baseline | 5 [4 to 5] | 5 [4 to 5] | 5 [4 to 5] | 5 [5 to 5]
  P[8]: Day 56: number analyzed (Participants) | 135 | 136 | 130 | 135
  P[8]: Day 56 | 6 [5 to 6] | 8 [6 to 9] | 8 [7 to 9] | 7 [6 to 9]
  P[8]: Day 84: number analyzed (Participants) | 130 | 129 | 130 | 131
  P[8]: Day 84 | 6 [5 to 7] | 11 [9 to 13] | 9 [8 to 11] | 8 [7 to 10]

8. Primary Outcome: Geometric Mean Titers of Neutralizing Antibody Against Rotavirus Strains Among Infants
Description: Neutralizing antibodies to each of the three rotavirus strains from which the vaccine antigens were derived (Wa, DS-1, and 1076) were measured at Baseline and 28 days after the second injection (Day 56 pre-vaccination; secondary outcome) and third injection (Day 84; primary outcome).
Time Frame: Baseline and Days 56 (pre-vaccination) and 84
Population: Per-protocol population participants with valid specimens at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 135 | 137 | 132 | 137
titer
  Strain Wa: Baseline | 118 [99 to 142] | 154 [131 to 181] | 128 [108 to 152] | 130 [110 to 153]
  Strain Wa: Day 56: number analyzed (Participants) | 135 | 137 | 131 | 136
  Strain Wa: Day 56 | 42 [34 to 52] | 90 [77 to 104] | 85 [74 to 97] | 85 [75 to 96]
  Strain Wa: Day 84: number analyzed (Participants) | 130 | 132 | 132 | 134
  Strain Wa: Day 84 | 42 [34 to 52] | 90 [77 to 104] | 85 [74 to 97] | 85 [75 to 96]
  Strain DS-1: Baseline | 54 [45 to 64] | 51 [41 to 62] | 44 [36 to 54] | 46 [38 to 57]
  Strain DS-1: Day 56: number analyzed (Participants) | 134 | 137 | 131 | 136
  Strain DS-1: Day 56 | 16 [13 to 19] | 26 [22 to 30] | 26 [22 to 31] | 27 [23 to 32]
  Strain DS-1: Day 84: number analyzed (Participants) | 130 | 131 | 132 | 134
  Strain DS-1: Day 84 | 11 [9 to 13] | 49 [42 to 58] | 48 [42 to 55] | 53 [46 to 61]
  Strain 1076: Baseline | 31 [25 to 38] | 37 [31 to 44] | 30 [25 to 36] | 35 [29 to 42]
  Strain 1076: Day 56: number analyzed (Participants) | 135 | 137 | 131 | 136
  Strain 1076: Day 56 | 12 [10 to 15] | 18 [16 to 22] | 18 [15 to 21] | 20 [17 to 23]
  Strain 1076: Day 84: number analyzed (Participants) | 130 | 132 | 132 | 134
  Strain 1076: Day 84 | 10 [8 to 11] | 34 [29 to 40] | 35 [30 to 40] | 43 [38 to 49]

9. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE) Over the Entire Study Period
Description: Any symptom starting after 7 days post any study injection was recorded as an adverse event. A serious adverse event (SAE) is any event that occurred from the first dose of study drug that resulted in any of the following outcomes:
  * Death - Life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Congenital abnormality or birth defect
  * Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant or require medical or surgical intervention to prevent one of the outcomes listed in the above definition of serious event.
  AEs related to study drug were those events for which there was a reasonable possibility that the study drug caused the event In the opinion of the site investigator.
Time Frame: Up to 6 months after the last injection (224 days for adults and infants; 168 days for toddlers)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8 | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12 | 139 | 139 | 140 | 139
Participants
  Any adverse event | 2 | 8 | 11 | 5 | 9 | 8 | 132 | 129 | 134 | 130
  Any serious adverse event | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 13 | 6 | 8
  Any grade 2 or higher AE | 0 | 2 | 1 | 0 | 2 | 2 | 27 | 43 | 28 | 36
  Any AE related to study drug | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 3 | 3
  Any grade 2 or higher AE related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

10. Secondary Outcome: Number of Infants With Anti-P2-VP8 Immunoglobulin G (IgG) Seroresponse 4 Weeks After the Second Vaccination, by Vaccine Antigen
Description: Seroresponse was defined as a four-fold rise or greater in antibody titer between Baseline and 28 days after the 2nd injection (Day 56). Measured by enzyme-linked immunosorbent assay (ELISA) and adjusted for decay in maternal antibodies. The estimated maternal antibody half-life was derived from linear regression of Log2 transformed titers in placebo recipients from the combined infant cohorts.
Time Frame: Day 56, pre-vaccination
Population: Per-protocol population; participants with available data for each antigen
Measure: Count of Participants; unit: Participants
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 135 | 137 | 131 | 136
Participants
  P[4] | 7 | 126 | 121 | 131
  P[6] | 25 | 136 | 125 | 133
  P[8]: number analyzed (Participants) | 134 | 137 | 131 | 136
  P[8] | 7 | 126 | 119 | 131
  Any 2 antigens | 7 | 126 | 121 | 132
  All 3 antigens: number analyzed (Participants) | 134 | 137 | 131 | 136
  All 3 antigens | 4 | 126 | 114 | 128

11. Secondary Outcome: Number of Infants With Anti-P2-VP8 Immunoglobulin A (IgA) Seroresponse 4 Weeks After the Second Vaccination, by Vaccine Antigen
Description: Seroresponse was defined as a four-fold rise or greater in antibody titer between Baseline and 28 days after the second injection (Day 56). Measured by enzyme-linked immunosorbent assay (ELISA) to whole viral lysate.
Time Frame: Day 56, pre-vaccination
Population: Per-protocol population; participants with available data for each antigen
Measure: Count of Participants; unit: Participants
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 135 | 137 | 131 | 136
Participants
  P[4]: number analyzed (Participants) | 134 | 136 | 131 | 136
  P[4] | 6 | 22 | 29 | 20
  P[6]: number analyzed (Participants) | 134 | 137 | 131 | 136
  P[6] | 12 | 22 | 33 | 27
  P[8]: number analyzed (Participants) | 135 | 136 | 130 | 135
  P[8] | 6 | 19 | 22 | 18
  Any 2 antigens: number analyzed (Participants) | 135 | 136 | 131 | 136
  Any 2 antigens | 7 | 19 | 25 | 21
  All 3 antigens: number analyzed (Participants) | 134 | 136 | 130 | 135
  All 3 antigens | 4 | 9 | 16 | 10

12. Secondary Outcome: Number of Infants With Neutralizing Antibody Responses 4 Weeks After the Second Vaccination
Description: Neutralizing antibody response was defined as a ≥ 2.7-fold rise in antibody titer between Baseline and 28 days after the second injection (Day 56). Neutralizing antibodies to each of the three rotavirus strains from which the vaccine antigens were derived (Wa, DS-1, and 1076) were measured using a validated assay. For infants, antibody titers were adjusted for decay in maternal antibodies.
Time Frame: Day 56, prevaccination
Population: Per-protocol population, participants with available data for each strain
Measure: Count of Participants; unit: Participants
Arm/Group | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 135 | 137 | 131 | 136
Participants
  Rotavirus strain Wa | 16 | 49 | 51 | 49
  Rotavirus strain DS-1: number analyzed (Participants) | 134 | 137 | 131 | 136
  Rotavirus strain DS-1 | 19 | 38 | 44 | 48
  Rotavirus strain 1076 | 13 | 29 | 33 | 32
  Any 2 strains | 14 | 35 | 38 | 37
  All 3 strains: number analyzed (Participants) | 134 | 137 | 131 | 136
  All 3 strains | 4 | 12 | 13 | 13

13. Secondary Outcome: Number of Adults and Toddlers With Anti-P2-VP8 Immunoglobulin G (IgG) Seroresponse, by Vaccine Antigen
Description: Seroresponse was defined as a four-fold rise or greater in IgG antibody titer between Baseline and 28 days after the final injection (Day 84 for adults and Day 28 for toddlers). Measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 84 for adults; Day 28 for toddlers
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
Participants
  P[4] | 0 | 11 | 11 | 0 | 7 | 11
  P[6] | 0 | 10 | 11 | 0 | 9 | 11
  P[8] | 0 | 11 | 11 | 0 | 10 | 10
  Any 2 antigens | 0 | 11 | 11 | 0 | 9 | 12
  All 3 antigens | 0 | 10 | 11 | 0 | 6 | 8

14. Secondary Outcome: Number of Adults and Toddlers With Anti-P2-VP8 Immunoglobulin A (IgA) Seroresponse, by Vaccine Antigen
Description: Seroresponse was defined as a four-fold rise or greater in IgA antibody titer between Baseline and 28 days after the final injection (Day 84 for adults and Day 28 for toddlers). Measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 84 for adults; Day 28 for toddlers
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
Participants
  P[4] | 0 | 11 | 11 | 0 | 8 | 11
  P[6] | 0 | 9 | 9 | 0 | 6 | 8
  P[8] | 0 | 11 | 10 | 0 | 10 | 10
  Any 2 antigens | 0 | 11 | 10 | 0 | 9 | 10
  All 3 antigens | 0 | 9 | 9 | 0 | 5 | 8

15. Secondary Outcome: Number of Adults and Toddlers With Neutralizing Antibody Responses to Each Rotavirus Strain
Description: Neutralizing antibody response was defined as a ≥ 2.7-fold rise in antibody titer between Baseline and 28 days after the final injection (Day 84 for adults and Day 28 for toddlers) for each of the three rotavirus strains from which the vaccine antigens were derived (Wa, DS-1, and 1076).
Time Frame: Day 84 for adults; Day 28 for toddlers
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
Participants
  Rotavirus strain Wa | 0 | 3 | 8 | 0 | 1 | 5
  Rotavirus strain DS-1 | 0 | 5 | 4 | 0 | 1 | 3
  Rotavirus strain 1076 | 0 | 2 | 3 | 0 | 0 | 2
  Any 2 strains | 0 | 3 | 3 | 0 | 0 | 2
  All 3 strains | 0 | 1 | 3 | 0 | 0 | 1

16. Secondary Outcome: Anti-P2-VP8 Immunoglobulin G (IgG) Geometric Mean Titers Among Adults and Toddlers, by Vaccine Antigen
Description: Measured at Baseline and 28 days after the final injection (Day 84 for adults; Day 28 for toddlers).
Time Frame: Baseline and Day 28 for toddlers or Day 84 for adults
Population: Per protocol population; participants with valid specimens at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12
titer
  P[4]: Baseline | 425 [198 to 909] | 358 [215 to 596] | 444 [314 to 627] | 183 [64 to 523] | 195 [89 to 425] | 282 [124 to 642]
  P[4]: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  P[4]: 28 days post-final vaccination | 311 [84 to 1156] | 11642 [7560 to 17927] | 13337 [8229 to 21616] | 174 [57 to 527] | 920 [285 to 2974] | 2396 [1089 to 5274]
  P[6]: Baseline | 89 [34 to 232] | 251 [90 to 695] | 234 [101 to 541] | 58 [20 to 165] | 172 [65 to 457] | 150 [86 to 262]
  P[6]: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  P[6]: 28 days post-final vaccination | 89 [14 to 576] | 22120 [12905 to 37916] | 29706 [17801 to 49573] | 72 [27 to 192] | 1767 [468 to 6672] | 2515 [884 to 7158]
  P[8]: Baseline | 140 [39 to 509] | 205 [109 to 387] | 220 [126 to 386] | 229 [70 to 751] | 113 [42 to 416] | 231 [73 to 731]
  P[8]: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  P[8]: 28 days post-final vaccination | 113 [24 to 529] | 11355 [7138 to 18063] | 14557 [8892 to 23831] | 294 [70 to 1239] | 1207 [389 to 3749] | 4059 [2022 to 8149]

17. Secondary Outcome: Anti-P2-VP8 Immunoglobulin A (IgA) Geometric Mean Titers Among Adults and Toddlers, by Vaccine Antigen
Description: Measured at Baseline and 28 days after the final injection (Day 84 for adults; Day 28 for toddlers).
Time Frame: Baseline and Day 28 for toddlers or Day 84 for adults
Population: Per-protocol population participants with valid specimens at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12
titer
  P[4]: Baseline | 151 [34 to 676] | 186 [78 to 445] | 143 [69 to 297] | 174 [32 to 936] | 124 [45 to 338] | 49 [18 to 135]
  P[4]: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  P[4]: 28 days post-final vaccination | 202 [15 to 2654] | 4685 [1395 to 15734] | 4533 [1990 to 10326] | 221 [55 to 897] | 629 [204 to 1935] | 443 [180 to 1091]
  P[6]: Baseline | 56 [25 to 127] | 120 [56 to 257] | 113 [43 to 296] | 16 [5 to 49] | 55 [22 to 137] | 15 [9 to 27]
  P[6]: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  P[6]: 28 days post-final vaccination | 95 [38 to 236] | 2470 [796 to 7659] | 1864 [505 to 6886] | 15 [4 to 65] | 198 [69 to 569] | 101 [37 to 274]
  P[8]: Baseline | 119 [23 to 614] | 151 [60 to 380] | 89 [40 to 201] | 136 [14 to 1294] | 83 [24 to 293] | 41 [13 to 131]
  P[8]: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  P[8]: 28 days post-final vaccination | 194 [19 to 2010] | 3590 [1060 to 12156] | 2350 [766 to 7210] | 211 [18 to 2480] | 928 [324 to 2653] | 530 [211 to 1333]

18. Secondary Outcome: Geometric Mean Titers of Neutralizing Antibody Against Rotavirus Strains Among Adults and Toddlers
Description: Measured at Baseline and 28 days after the final injection (Day 84 for adults; Day 28 for toddlers).
Time Frame: Baseline and Day 28 for toddlers or Day 84 for adults
Population: Per-protocol population participants with valid specimens at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 12 | 12
titer
  Strain Wa: Baseline | 317 [123 to 820] | 448 [247 to 815] | 276 [193 to 396] | 77 [16 to 369] | 131 [46 to 373] | 67 [25 to 176]
  Strain Wa: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  Strain Wa: 28 days post-final vaccination | 244 [80 to 743] | 913 [579 to 1439] | 815 [531 to 1251] | 78 [16 to 370] | 147 [47 to 459] | 253 [119 to 537]
  Strain DS-1: Baseline | 76 [16 to 355] | 114 [57 to 228] | 119 [57 to 248] | 16 [3 to 85] | 29 [9 to 92] | 20 [9 to 44]
  Strain DS-1: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  Strain DS-1: 28 days post-final vaccination | 59 [4 to 813] | 390 [278 to 545] | 317 [152 to 659] | 15 [3 to 79] | 40 [14 to 113] | 60 [22 to 167]
  Strain 1076: Baseline | 77 [14 to 415] | 175 [74 to 416] | 152 [63 to 366] | 13 [3 to 53] | 28 [9 to 89] | 16 [8 to 34]
  Strain 1076: 28 days post-final vaccination: number analyzed (Participants) | 4 | 11 | 11 | 6 | 12 | 12
  Strain 1076: 28 days post-final vaccination | 43 [4 to 428] | 354 [180 to 695] | 284 [132 to 607] | 15 [3 to 67] | 30 [9 to 99] | 25 [11 to 58]

19. Post Hoc Outcome: Number of Adults and Infants With ≥ 4-fold Rise in Neutralizing Antibody Titer to Each Rotavirus Strain
Description: The number of adults and infants with a 4-fold or greater increase from Baseline in neutralizing antibody titers to each of the three rotavirus strains from which the vaccine antigens were derived 4 weeks after the second (Day 56) and third (Day 84) vaccinations.
  For infants, antibody titer was adjusted for decay in maternal antibodies.
Time Frame: Day 56 and Day 84
Population: Per-protocol population participants with valid specimens at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: Placebo | Adults: 30 µg P2-VP8 | Adults: 90 µg P2-VP8 | Infants: Placebo | Infants: 15 µg P2-VP8 | Infants: 30 µg P2-VP8 | Infants: 90 µg P2-VP8
Number analyzed (Participants) | 4 | 11 | 11 | 135 | 137 | 132 | 136
Participants
  Strain Wa: Day 56: number analyzed (Participants) | 4 | 11 | 11 | 135 | 137 | 131 | 136
  Strain Wa: Day 56 | 0 | 0 | 4 | 9 | 31 | 29 | 23
  Strain Wa: Day 84: number analyzed (Participants) | 4 | 11 | 11 | 130 | 132 | 132 | 134
  Strain Wa: Day 84 | 0 | 2 | 3 | 17 | 73 | 95 | 92
  Strain DS-1: Day 56: number analyzed (Participants) | 4 | 11 | 11 | 134 | 137 | 131 | 136
  Strain DS-1: Day 56 | 0 | 5 | 2 | 11 | 25 | 30 | 30
  Strain DS-1: Day 84: number analyzed (Participants) | 4 | 11 | 11 | 130 | 131 | 132 | 134
  Strain DS-1: Day 84 | 0 | 4 | 4 | 17 | 85 | 96 | 93
  Strain 1076: Day 56: number analyzed (Participants) | 4 | 11 | 11 | 135 | 137 | 131 | 136
  Strain 1076: Day 56 | 0 | 1 | 1 | 7 | 21 | 20 | 18
  Strain 1076: Day 84: number analyzed (Participants) | 4 | 11 | 11 | 130 | 132 | 132 | 134
  Strain 1076: Day 84 | 0 | 2 | 3 | 13 | 73 | 86 | 98

20. Post Hoc Outcome: Number of Toddlers With ≥ 4-fold Rise in Neutralizing Antibody Titer to Each Rotavirus Strain
Description: The number of toddlers with a 4-fold or greater increase from Baseline 4 weeks after vaccination in neutralizing antibody titers to each of the three rotavirus strains from which the vaccine antigens were derived.
Time Frame: Day 28
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Toddlers: Placebo | Toddlers: 30 µg P2-VP8 | Toddlers: 90 µg P2-VP8
Number analyzed (Participants) | 6 | 12 | 12
Participants
  Rotavirus strain Wa | 0 | 0 | 4
  Rotavirus strain DS-1 | 0 | 1 | 3
  Rotavirus strain 1076 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months after the last injection (224 days for adults and infants; 168 days for toddlers)
Arm/Group | Adult: Placebo | Adult: P2-VP8 (30 µg) | Adult: P2-VP8 (90 µg) | Toddler: Placebo | Toddler: P2-VP8 (30 µg) | Toddler: P2-VP8 (90 µg) | Infant: Placebo | Infant: P2-VP8 (15 µg) | Infant: P2-VP8 (30 µg) | Infant: P2-VP8 (90 µg)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/12 | 0/6 | 0/12 | 0/12 | 1/139 | 1/140 | 1/140 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12 | 0/12 | 0/6 | 1/12 | 1/12 | 8/139 | 13/139 | 6/140 | 8/139
Other Adverse Events (participants affected / at risk) | 2/6 | 8/12 | 11/12 | 5/6 | 9/12 | 8/12 | 132/139 | 129/139 | 134/140 | 130/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult: Placebo (N=6) | Adult: P2-VP8 (30 µg) (N=12) | Adult: P2-VP8 (90 µg) (N=12) | Toddler: Placebo (N=6) | Toddler: P2-VP8 (30 µg) (N=12) | Toddler: P2-VP8 (90 µg) (N=12) | Infant: Placebo (N=139) | Infant: P2-VP8 (15 µg) (N=139) | Infant: P2-VP8 (30 µg) (N=140) | Infant: P2-VP8 (90 µg) (N=139)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult: Placebo (N=6) | Adult: P2-VP8 (30 µg) (N=12) | Adult: P2-VP8 (90 µg) (N=12) | Toddler: Placebo (N=6) | Toddler: P2-VP8 (30 µg) (N=12) | Toddler: P2-VP8 (90 µg) (N=12) | Infant: Placebo (N=139) | Infant: P2-VP8 (15 µg) (N=139) | Infant: P2-VP8 (30 µg) (N=140) | Infant: P2-VP8 (90 µg) (N=139)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 4 | 12 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 26 | 15 | 16 | 22
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 6 | 1 | 2
Influenza like illness (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 5 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 13 | 22 | 20 | 19
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida nappy rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 4
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 15 | 8 | 10 | 14
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 3 | 8
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 16 | 10 | 15
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 12 | 10 | 8 | 8
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 10 | 9 | 15
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 4 | 3
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 1
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 5 | 3
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Respiratory syncytial virus bronchiolitis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 22 | 27 | 29
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tinea faciei (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 6 | 2 | 4 | 5 | 70 | 84 | 74 | 82
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaccination site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Penile swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 9 | 11 | 17 | 15
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 28 | 34 | 24 | 47
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 20 | 15 | 12 | 19
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 5
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 10 | 14 | 14
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 13 | 10 | 17
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 2
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT02646891/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT02646891/SAP_001.pdf